CLINICAL TRIAL: NCT01967160
Title: A Non-interventional Pharmacovigilance Study of Osteonecrosis of the Jaw and Infection Leading to Hospitalization Among Patients With Cancer Treated With XGEVA™ or Zoledronic Acid in Sweden, Denmark, and Norway
Brief Title: Osteonecrosis of the Jaw (ONJ) and Infection Among Nordic Cancer Patients Treated With XGEVA™ or Zoledronic Acid
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20101363
Record Dates: First submitted 2013-10-18; First posted 2013-10-22 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2021-09

CONDITIONS: Osteonecrosis of the Jaw; Infection Leading to Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- XGEVA inception cohort: Patients with cancer who are naïve to oral or IV bisphosphonate treatment at the dose indicated for SRE prevention and who begin treatment with XGEVA at any time during the treatment cohort identification period
- Zoledronic acid inception cohort: Patients with cancer who are naïve to oral or IV bisphosphonate treatment at the dose indicated for SRE prevention and who begin treatment with IV zoledronic acid at any time during the treatment cohort identification period
- XGEVA-switch cohort: Patients with cancer who switch to XGEVA during treatment cohort identification period after having started antiresorptive therapy at the dose indicated for SRE prevention of no more than 2 years duration with bisphosphonates (<24 IV infusions or <24 monthly oral prescriptions)

SUMMARY:
A non-interventional study to assess incident rates of Osteonecrosis of the Jaw and Infections leading to hospitalization in Cancer patients treated with XGEVA™ in Sweden, Denmark and Norway.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* diagnosed with cancer
* subsequent to cancer diagnosis, initiating cancer-related antiresorptive treatment during the treatment cohort identification period with XGEVA or zoledronic acid or switching to XGEVA from cancer-related treatment with oral or IV bisphosphonates at the dose indicated for SRE prevention of less than 2 years duration (≤ 24 IV infusions or ≤ 24 monthly oral prescriptions)

Exclusion Criteria:

* history of radiation treatment for head and neck cancer before a subject's potential index date
* hypercalcemia of malignancy as the sole indication for treatment with an anti-resorptive agent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients treated with antiresorptive therapies for SRE prevention
Sampling Method: Probability Sample
Enrollment: 2560 (Actual)
Dates: Start 2012-01-02 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
1. Incidence proportions of medically confirmed osteonecrosis of the jaw (ONJ) in XGEVA and zoledronic acid inception cohorts | 5 years
2. Incidence proportions of infections leading to hospitalization in XGEVA and zoledronic acid inception cohorts | 3 years

SECONDARY OUTCOMES:
1. Incidence proportions of medically confirmed ONJ in the cohort switching from an oral or IV bisphosphonate (at the dose indicated for cancer patients to prevent skeletal related events) to XGEVA | 5 years
2. Incidence proportions of medically confirmed ONJ in the cohort switching from an oral or IV bisphosphonate (at the dose indicated for cancer patients to prevent SREs) to XGEVA stratified by number of prior cancer-related bisphosphonate treatments | 5 years
3. Characterize the XGEVA inception, zoledronic acid inception, and the XGEVA-switch cohorts with respect to patient characteristics, cancer type, medical history, and number of bisphosphonate or XGEVA treatments at the dose indicated for SRE prevention | 5 years
4. Summarize oral risk factor information for medically confirmed ONJ cases | 5 years
5. Summarize for medically confirmed ONJ cases information on ONJ stage, treatment, clinical course, and resolution | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Acquavella J, Ehrenstein V, Schiodt M, Heide-Jorgensen U, Kjellman A, Hansen S, Larsson Wexell C, Herlofson BB, Noerholt SE, Ma H, Ohrling K, Hernandez RK, Sorensen HT. Design and methods for a Scandinavian pharmacovigilance study of osteonecrosis of the jaw and serious infections among cancer patients treated with antiresorptive agents for the prevention of skeletal-related events. Clin Epidemiol. 2016 Jul 20;8:267-72. doi: 10.2147/CLEP.S107270. eCollection 2016. PMID 27499646
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com